CLINICAL TRIAL: NCT07091617
Title: AYA Access Study: An Enhanced eHealth and Chat-Bot Enabled Delivery Model for Clinical Genetic Services in Community AYA Cancer Patients
Brief Title: Testing an Enhanced Digital Delivery Model for Inherited Cancer Genetic Testing in Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A232301CD; NCI-2025-02152 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2025-06-24; First posted 2025-07-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Miscellaneous Neoplasm, Nos; Non-Neoplastic Condition, Nos
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — Telemedicine; Genetic Testing; Early Intervention, Educational; Patient Navigation; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard remote genetic services) (Active Comparator): Patients attend a standard of care telehealth visit with a genetic counselor for pretest genetic education. Patients then undergo standard of care genetic testing and attend a telehealth visit with a genetic counselor for disclosure of results.
  Interventions: Other: Telemedicine; Other: Genetic Testing; Other: Survey Administration
- Arm II (Genetic Journey Chatbot) (Experimental): Patients receive access to the Genetic Journey Chatbot and choose to complete digital pre-test genetic education via the digital tool or via telehealth visit with a genetic counselor. Via the chatbot, patients may request a telehealth visit with a genetic counselor at any time to answer unresolved questions. Patients then undergo standard of care genetic testing and attend a telehealth visit with a genetic counselor for disclosure of results. The chatbot remains available to answer questions, assess barriers, and provide reminders for next steps during the testing period.
  Interventions: Other: Telemedicine; Other: Genetic Testing; Other: Internet-Based Intervention; Other: Educational Intervention; Behavioral: Patient Navigation; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Telemedicine — Undergo telehealth visit with genetic counselor for pretest genetic education
Other: Genetic Testing — Complete standard of care genetic testing
Other: Telemedicine — Undergo telehealth visit with genetic counselor for disclosure of results
Other: Internet-Based Intervention — Receive access to Genetic Journey Chatbot
  Arms: Arm II (Genetic Journey Chatbot)
Other: Educational Intervention — Complete digital pre-test genetic education
  Arms: Arm II (Genetic Journey Chatbot)
Behavioral: Patient Navigation — Utilize chatbot to answer questions, assess barriers, and provide reminders for next steps during the testing period
  Arms: Arm II (Genetic Journey Chatbot)
Other: Interview — Complete interview
  Arms: Arm II (Genetic Journey Chatbot)
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase III trial compares the use of a digital chatbot enabled intervention to standard remote genetic services for increasing uptake of genetic counseling and testing among adolescents and young adult (AYA) cancer patients. Genetic testing for cancer predisposition syndromes has become standard evidence-based practice and can inform enhanced screening and risk reducing measures to reduce cancer morbidity and mortality. Despite this, many AYAs are not receiving recommended genetic counseling and testing. Offering remote telehealth services can address access barriers and chatbots and texting interventions could enhance patient outcomes and reduce provider and staff time. The use of a digital chatbot enabled intervention may be equally as effective as standard remote genetic services in AYA cancer patients undergoing genetic testing.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To evaluate the efficacy of an enhanced eHealth and chatbot enabled delivery model to increase uptake of genetic counseling.

II. To evaluate the efficacy of an enhanced eHealth and chatbot enabled delivery model to increase uptake of genetic testing.

SECONDARY OBJECTIVE:

I. To evaluate the efficacy of an enhanced eHealth and chatbot enabled delivery model to provide non-inferior short-term and longitudinal cognitive (e.g. knowledge), affective (e.g. distress), and behavioral outcomes (e.g. cancer screening and communication to relatives) and costs.

EXPLORATORY OBJECTIVES:

I. To test for moderators of uptake of counseling and testing (primary objectives).

II. To test for moderators of short-term and longitudinal patient outcomes (secondary objectives).

III. To identify facilitators and barriers to implementation of the enhanced eHealth and chatbot enabled delivery model and standard remote services.

OUTLINE: Patients are randomized to 1 of 2 arms. Non-patient participants are assigned to arm 3.

ARM I: Patients attend a standard of care telehealth visit with a genetic counselor for pretest genetic education. Patients then undergo standard of care genetic testing and attend a telehealth visit with a genetic counselor for disclosure of results.

ARM II: Patients receive access to the Genetic Journey Chatbot and choose to complete digital pre-test genetic education via the digital tool or via telehealth visit with a genetic counselor. Via the chatbot, patients may request a telehealth visit with a genetic counselor at any time to answer unresolved questions. Patients then undergo standard of care genetic testing and attend a telehealth visit with a genetic counselor for disclosure of results. The chatbot remains available to answer questions, assess barriers, and provide reminders for next steps during the testing period.

ARM III: Non-patient participants complete an interview on study.

After completion of study intervention, patients are followed up at 6 and 12 months.

ELIGIBILITY:
* PATIENTS: Age ≥ 18 years and ≤ 39 years at the time of enrollment
* PATIENTS: AYA cancer patients and survivors. This includes patients at any stage of diagnosis (e.g., newly diagnosed, in treatment, in survivorship) and a cancer diagnosis (including pediatric cancers) at any age ≤ 39 years old. Given targeted therapies for BRCA+ and microsatellite instability (MSI)-high/Lynch Syndrome patients and benefit to relatives, patients with metastatic cancer are included. Any history of cancer, regardless of being in treatment or not
* PATIENTS: Language: In order to complete the mandatory patient-completed measures and receive genetic education and counseling, participants must be able to speak and read English or Spanish
* PATIENTS: No known diagnosis of dementia or cognitive impairment. Persons with impaired decision-making capacity are ineligible as they need to be able to understand genetic test results, its implications for the patient and family, and explain genetic test results to their family members
* PATIENTS: No persons with a known psychiatric or documented developmental disorder that affects cognitive or emotional functions to the extent that the capacity for judgment and reason is significantly diminished, such that they cannot participate based on the judgment of the treating physician
* PATIENTS: Participants must meet National Comprehensive Cancer Network (NCCN) guidelines for genetic testing assessment provided by Penn Telegenetics by the Eligibility Verification Assessment (EVA) chatbot, or paper forms and genetic counselor's review
* NON-PATIENT PARTICIPANT: Non-patient participants eligible for this study include: oncology providers, members of the care team and clinic staff, genetic counselors, and insurers (i.e., people who work in financial services and/or for insurance companies) who participate in oncology care among AYA in community for this study
* NON-PATIENT PARTICIPANT: Age ≥ 18 years
* NON-PATIENT PARTICIPANT: Non-patient participants must be able to speak and read English or Spanish in order to participate in the key informant interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 535 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2030-11-23 (Estimated); Study Completion 2031-01-15 (Estimated)

PRIMARY OUTCOMES:
Uptake of genetic counseling | Within 6 months of baseline
  Defined as a binary outcome of whether an adolescent or young adult (AYA) underwent genetic counseling within 6 months post completion of the baseline survey. Will be compared between randomized arms using Cochran-Mantel-Haenszel (CMH) tests stratified by gender and a Bonferroni correction will be applied to control family-wise type I error.
Uptake of genetic testing | Within 6 months of baseline
  Defined as a binary outcome of whether an AYA underwent genetic testing within 6 months post completion of the baseline survey. Will be compared between randomized arms using CMH tests stratified by gender and a Bonferroni correction will be applied to control family-wise type I error.

SECONDARY OUTCOMES:
Knowledge of genetic disease | Up to 42 months post registration
  Obtained from the KnowGene scale. Will be compared using non-inferiority testing with the equivalent of a 0.3 standard deviation (SD) non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Test result recall | Up to 42 months post registration
  Measured via the Test Result Recall scale. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for each secondary endpoint at T2 (the primary time point of interest for the secondary analyses) will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Perceptions of genetic disease | Up to 42 months post registration
  Measured via the Perceived Risk scale. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Anxiety | Up to 42 months post registration
  Measured via Patient Reported Outcome Measurement Information System (PROMIS) anxiety score. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Depression | Up to 42 months post registration
  Measured via PROMIS Depression score. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Disease-specific distress | Up to 42 months post registration
  Measured via the Revised Impact of Events Scale score. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Impact of cancer risk | Up to 42 months post registration
  Measured via the Multi-dimensional Impact of Cancer Risk Assessment score. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit or each secondary endpoint at T2 (the primary time point of interest for the secondary analyses) will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics
Satisfaction with genetic services | Up to 30 months post registration
  Measured via the Satisfaction with Genetic Services scale. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit or each secondary endpoint at T2 (the primary time point of interest for the secondary analyses) will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD.
Attitude toward genetic testing | Up to 24 months post registration
  Measured via Attitudes Toward Genetic Testing scale. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit or each secondary endpoint at T2 (the primary time point of interest for the secondary analyses) will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD.
Lifestyle behaviors | Up to 42 months post registration
  Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Health behaviors | Up to 42 months post registration
  Measured via the Screening Health behaviors score. Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Communication to at-risk relatives | Up to 42 months post registration
  Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Genetic counselor time | Up to 24 months post registration
  o Will be compared using non-inferiority testing with the equivalent of a 0.3 SD non-inferiority margin. The lower limit of the one-sided 97.5% confidence limit for the difference in means will be compared with the non-inferiority margin and non-inferiority will be concluded if the interval fully lies above -0.3 SD. Longitudinal analyses will include model based analysis using generalized linear models of endpoints over time with link function determined by distribution of the endpoint being modeled and adjusting for baseline patient and disease characteristics.
Testing costs | Up to 36 months post registration
  Measured by 2 patient reported items
Costs of the intervention | Up to 42 months post registration
  o Will be estimated from a societal perspective, including direct medical and nonmedical costs. These include intervention and chatbot hosting, telecommunication services, personnel and patient time. Information to estimate intervention costs collected from study billing and payment records (e.g. website hosting, chatbot usage and time, videoconferencing and phone usage) and telegenetic staff logs (personnel time). The cost of personnel time will be based on institution-specific salaries, including fringe benefits. In sensitivity analysis, will substitute site-specific salary information with national average wage rates for the relevant occupational categories. Information about other out-of-pocket costs for testing (e.g. copayments) will be obtained through participant surveys. Patient time costs will be valued using national average wage rates for participant-specified occupations.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bradbury, MD, Study Chair — Alliance for Clinical Trials in Oncology
Locations (201):
- United States (201):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Mercy Cancer Center, Merced, California
  - Providence Queen of The Valley, Napa, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Saint Joseph's Medical Center, Stockton, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided